CLINICAL TRIAL: NCT02144805
Title: Evaluation of Single Versus Double-layer Technique by Closure of Cesarean Uterine Incision. A Randomized Controlled Study
Brief Title: Closure of Uterine Incision by Single or Double Layer Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-29
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Pregnancy
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suturing in a single layer (Active Comparator): The technique used for single layer to close the uterine incision following cesarean sectio
  Interventions: Procedure: Suturing in a single layer
- Suturing in two layer (Active Comparator): The technique used for two layer technie to close the uterine incision following cesarean sectio
  Interventions: Procedure: Suturing in two layer

INTERVENTIONS:
Procedure: Suturing in a single layer — The procedure define the use of one single suture for closure of the uterine incision following cesarean section.
  Arms: Suturing in a single layer
Procedure: Suturing in two layer — The procedure define the use of two sutures for closing the uterine incision following cesarean section
  Arms: Suturing in two layer

SUMMARY:
The study compares short-term and long-term effects on myometrial thickness in women sutured by single- or double-layer technique by closure of cesarean uterine incision. The study is a randomized clinically controlled study.

DETAILED DESCRIPTION:
Objective: To compare short-term and long-term effects on myometrial thickness in women sutured by single- or double-layer technique by closure of cesarean uterine incision. The study is a randomized clinically controlled study.

Design:Follow-up by ultra sound of a randomised controlled trial. Surgical technique was blinded for the investigator.

Setting: An obstetric department in a tertiary referral hospital, 2008-2013. Participants: Healthy nulliparous scheduled for elective caesarean section randomly assigned to closure of the uterine incision by single- or double layer techniques.

Intervention: A modified version of the Misgav-Ladach surgical technique was used. The women were examined by abdominal ultra sound before discharge from the maternity ward, and by vaginal ultra sound and hysterosonography minimum five month post partum.

Main outcome measure: Thickness of the remaining myometrium corresponding to the former cesarean uterine incision measured by ultra sound.

ELIGIBILITY:
Inclusion Criteria:

* Women submitted to cesarean sectio

Exclusion Criteria:

* Exclusion criteria were: Former uterine operations such as myomectomy or surgery resulting in entering the cavity, fibroids located in the cervix or the cervicalcorporal border, inflammatory bowel disease, SLE, rheumatoid arthritis, IDDM, re-operations after inclusion or the cesarean section and more than three additional single sutures for hemostasis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Myometrial thickness | 5 months
  Thickness of the remaining myometrium corresponding to the former cesarean uterine incision measured by ultra sound

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Bennich, consultant, Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Roskilde, Roskilde, Denmark